CLINICAL TRIAL: NCT03117179
Title: Patient Follow-up After Consultation in Emergency Department
Acronym: APCSU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2013_843_0012
Record Dates: First submitted 2017-04-05; First posted 2017-04-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Consultation; Emergency
MeSH Terms: conditions — Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with an interview (Other)
  Interventions: Other: Discharge from patient after consultation in emergency department
- Patient without an interview (Other)
  Interventions: Other: Discharge from patient after consultation in emergency department

INTERVENTIONS:
Other: Discharge from patient after consultation in emergency department — Discharge from patient after consultation in emergency department

SUMMARY:
Each year more than 15 million French people visit the emergency services and almost 80% of them come out without hospitalization after having undergone a clinical examination and possibly additional examinations.

DETAILED DESCRIPTION:
Each year more than 15 million French people visit the emergency services and almost 80% of them come out without hospitalization after having undergone a clinical examination and possibly additional examinations.

Following their discharge, compliance with discharge requirements and recommendations (treatment, monitoring, follow-up, etc.) is a determining factor in improving their health. Non-membership is linked to an increase in morbidity, mortality and use of the health system. Patient adherence to discharge instructions is conditional on patient understanding. Unfortunately, the environment of an emergency service often creates conditions for information and education of the patient that are often far from optimal or at least that are specific to a typical consultation.

Data from the international literature showed that 78% of people who come out of emergency after consultation do not clearly understand the instructions and only 20% are aware of their lack of understanding. Waisman et al. Documented that 25% of patients did not understand their diagnosis and that 13% to 18% did not understand treatment instructions. Heng et al. Have shown that patients leaving after head trauma are unable to cite the symptoms that should prompt them to consult quickly.

The involvement of healthcare teams to inform patients with the help of different communication media is therefore particularly important in trying to improve understanding and adherence to exit instructions. However, Zavala et al. Point to the fact that this is not necessarily sufficient.

Some authors have identified factors of poor adherence: multiple chronic diseases, multiple drug treatments, psychiatric disorders, but also age, social isolation, depression, quality of life and socio-economic and cultural level , A low level of health literacy, or planned medical follow-up, the severity of the pathology and the perception of that severity by the patient, or the patient's dissatisfaction with medical instructions.

The patients' adherence to the literature is evaluated in a varied manner according to the pathologies concerned: counting the number of tablets; Patient self-tracking log; Reports from physicians, reports by third parties (such as the patient's spouse); Electronic measurements (for example, metered-dose inhalers or electronic drop dispensers); Blood or urine dosage. The different methods used have advantages and disadvantages that need to be assessed according to the needs of the study we wish to implement. While declarative investigations in the assessment of patient adherence are criticized, no method has unfortunately been used as a benchmark for assessing adherence. The bibliographic search did not find any questionnaires that had been validated in this context. In order to evaluate the adhesion, the investigator will therefore opt for a semi-directed interview at D7 in order to better control a possible bias of memorization. This tool has known limitations including a tendency to overestimate adhesion, because patients tend to respond to what doctors want to hear. This will be taken into account in the interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

* Major patient not benefiting from any legal protection measures.
* Speaking French.
* Outgoing after having received a consultation in a hospital emergency department.
* Accepting to participate in the study after being informed of the protocol.
* Having the possibility to be reached by telephone on J7.

Exclusion Criteria:

* Patient with a pathology that does not allow him or her to understand instructions or express themselves.
* Patient under tutelage or curatorship or deprived of all freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Analysis of patient compliance with discharge | 7 days
  Analysis of patient compliance with discharge orders issued after consultation in emergencies determined by telephone interview

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Result] Gignon M, Ammirati C, Mercier R, Detave M. Compliance with emergency department discharge instructions. J Emerg Nurs. 2014 Jan;40(1):51-5. doi: 10.1016/j.jen.2012.10.004. Epub 2013 Jan 7. PMID 23305946